CLINICAL TRIAL: NCT02875691
Title: The Effect of Green Tea Extract on Some Inflammatory Biomarkers(IL 6, IL1β,TNF α,CRP), Serum Total Antioxidant Capacity(TAC), MDA and Disease Activity in Patients With Systemic Lupus Erythematous
Brief Title: Effect of Green Tea on Treatment of Lupus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, zahra shamekhi, zahra shamekhi , phd student in Ahvaz Jundishapur University of Medical Sciences, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IR.AJUMS.REC.1394.251; IR.AJUMS.REC.1394.251 (Other: Ahvaz Jundishapur University of Medical Sciences)
Record Dates: First submitted 2016-05-28; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-05

CONDITIONS: Autoimmune; Lupus Erythematosus, Systemic
Keywords: disease activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- green tea extract (Active Comparator): Patients were given daily dose of 1000mg aqueous green tea extract (of 6 grams of dried green tea leaf) in the form of 2 capsules (500 mg) for three months.
  Interventions: Dietary Supplement: green tea extract
- Placebo (Placebo Comparator): Patients in placebo group received daily dose of 1000 mg cellulose in the form of 2 capsules (500 mg) for three months
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: green tea extract — Patients are given daily dose of 1000mg aqueous green tea extract (of 6 grams of dried green tea leaf) in the form of 2 capsules( 500 mg) for three months.
  Arms: green tea extract
Dietary Supplement: placebo — Patients in placebo group receive daily dose of 1000 mg cellulose in the form of 2 capsules (500 mg) for three months
  Arms: Placebo

SUMMARY:
This randomized double blind clinical trial performed on 68 patients (32 in intervention and 36 in control group) diagnosed with SLE. The patients in intervention group were given daily dose of 1000mg of aqueous green tea extract (of 6 gram of dried green tea leaf) in form of two capsules ( 500 mg). Also in control group, the patients were given daily dose of 1000mg of cellulose in form of two capsules ( 500 mg) Variables include SLE disease activity, some biomarkers of inflammation and oxidative stress and anthropometric indicators at baseline and end of the study.

The investigators used SLEDAI (systemic lupus erythematous disease activity index ) questionnaire for evaluating the clinical signs of the disease. The questionnaires filled out at baseline and after 3 month.

DETAILED DESCRIPTION:
noting

ELIGIBILITY:
Inclusion Criteria:

The patients older than 15 years,diagnosed with systemic lupus erythematous (SLE) according to ACR(American College of Rheumatology) criteria.

Exclusion Criteria:

* Patients with other autoimmune diseases (diabetes, ...)
* Cardiovascular disease
* Patients with infectious or liver disease;
* severe infection
* Pregnancy
* Breastfeeding
* Smoking
* Alcohol consumption
* Use of any dietary supplements
* Changing of medication during the study period

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
systemic lupus erythematous Disease Activity | Three months after starting of intervention
  Clinical signs consist of 24 items, 16 of which are clinical items such as seizure, psychosis, organic brain syndrome, visual disturbance, other neurological problems, hair loss, new rash, muscle weakness, arthritis, blood vessel inflammation, mouth sores, chest pain worse with deep breathing and manifestations of pleurisy and/or pericarditis and fever consistency.Eight of the 24 items are laboratory results such as urinalysis testing, blood complement levels, increase anti-DNA antibody levels, low platelets, and low white blood cell count. these items assessed by SLEDAI questionnaire

SECONDARY OUTCOMES:
measurement of some proinflammatory and anthropometric markers | At baseline and after three months of intervention
  interleukin-6 (IL6), interleukin1β(IL1β , Tumor Necrosis Factor-α (TNF-α),Total Antioxidant Capacity (TAC) of Blood serum will be assessed by enzyme-linked immunosorbent assay (ELISA) at baseline and after three months intervention
  • Malondialdehyde (MDA) Blood serum MDA will be assessed by Thiobarbituric acid method (TBA)
Health-Related Quality of Life | At baseline and after three months of intervention
  Quality of Life will be assessed by12-item Short-Form (SF-12v2) self-report questionnaire ,at baseline and after3 months of intervention

OTHER OUTCOMES:
Dietary intake | at baseline and after 3 month of intervention
  24-Hour dietary recalls questionnaires will be used to assess dietary pattern
Weight | at baseline and after 3 month of intervention
  Weight will be measured in kg
BMI | at baseline and after 3 month of intervention
  BMI is weight in kilograms divided to height in meters squared

CONTACTS AND LOCATIONS:
Overall Officials: Iran Ahvaz, Principal Investigator — Ahvaz University of Medical Sceinces, Ahvaz, Iran
Locations (1):
- Iran, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Undecided